CLINICAL TRIAL: NCT06989112
Title: DESTINY-Endometrial01: An Open-Label, Sponsor-Blinded, Randomized, Controlled, Multicenter, Phase III Study of Trastuzumab Deruxtecan (T-DXd) Plus Rilvegostomig or Pembrolizumab vs Chemotherapy Plus Pembrolizumab as First-Line Therapy of HER2-Expressing (IHC 3+/2+), Mismatch Repair Proficient (pMMR), Primary Advanced or Recurrent Endometrial Cancer
Brief Title: DESTINY-Endometrial01: A Phase III Study of Trastuzumab Deruxtecan Plus Rilvegostomig or Pembrolizumab as First-Line Treatment of HER2-Expressing (IHC 3+/2+), Mismatch Repair Proficient (pMMR) Endometrial Cancer
Acronym: DE-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Gynecologic Oncology Group (GOG) Foundation Inc. (Unknown); European Network for Gynaecological Oncological Trial groups(ENGOT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D781DC00001; 2023-508056-19-00 (Registry Identifier: CTIS (EU)); GOG-3098 (Other: Gynecologic Oncology Group Foundation); ENGOT-EN24 (Other: European Network for Gynaecological Oncological Trial groups)
Record Dates: First submitted 2025-03-11; First posted 2025-05-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Uterine Cancer; Endometrial Carcinoma; Human epidermal growth factor receptor 2 (HER2); PMMR; Trastuzumab deruxtecan; T-DXd; DS-8201a; Anti-HER2-Antibody Drug Conjugate(ADC); DESTINY-Endometrial01; Programmed Cell Death-1 (PD1, PD-1); Immune checkpoint inhibitor; TIGIT; Pembrolizumab; Carboplatin; Paclitaxel; Rilvegostomig
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — trastuzumab deruxtecan; pembrolizumab; Carboplatin; Paclitaxel; Docetaxel

STUDY DESIGN:
Intervention Model Description: Participants with HER2-expressing (IHC 3+/2+), pMMR, primary advanced (Stage III/IV) or recurrent EC will be randomly assigned to treatment with trastuzumab deruxtecan (T-DXd) plus rilvegostomig (Arm A), T-DXd plus pembrolizumab (Arm B), or chemotherapy (carboplatin plus paclitaxel) plus pembrolizumab (Arm C).
Masking Description: This is an open-label, Sponsor-blinded study. To maintain the integrity of the study, Sponsor personnel directly involved in study conduct will not undertake or have access to efficacy data aggregated by treatment arm prior to final data readout for the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: T-DXd + Rilvegostomig (Experimental): T-DXd IV Q3W plus rilvegostomig IV Q3W. Treatment will continue until objective disease progression according to RECIST v1.1 as assessed by the Investigator and confirmed by BICR or until other discontinuation criteria is met, whichever occurs first.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Rilvegostomig
- Arm B: T-DXd + Pembrolizumab (Experimental): T-DXd IV Q3W plus pembrolizumab IV Q3W. Treatment will continue until objective disease progression according to RECIST v1.1 as assessed by the Investigator and confirmed by BICR or until other discontinuation criteria is met, whichever occurs first.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Pembrolizumab
- Arm C: Carboplatin + Paclitaxel + Pembrolizumab (Active Comparator): Carboplatin, paclitaxel and pembrolizumab administered Q3W during 6 cycles, followed by maintenance with pembrolizumab IV Q6W during 14 cycles. Treatment with pembrolizumab will continue for up to 20 total cycles (approximately 24 months, accounting for combination and maintenance phases) or until other discontinuation criteria is met, whichever occurs first. At the discretion of the investigator, participants may continue to receive carboplatin, paclitaxel and pembrolizumab Q3W for up to 10 cycles. Docetaxel can be used as an alternative to paclitaxel for participants who had a hypersensitivity reaction to paclitaxel with a failed rechallenge (or not amenable to rechallenge), according to the investigator's clinical judgment.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Experimental therapy by intravenous infusion
  Other Names: DS-8201a, T-DXd
  Arms: Arm A: T-DXd + Rilvegostomig; Arm B: T-DXd + Pembrolizumab
Drug: Rilvegostomig — Experimental therapy by intravenous infusion
  Arms: Arm A: T-DXd + Rilvegostomig
Drug: Pembrolizumab — Immunotherapy by intravenous infusion
  Other Names: Keytruda
  Arms: Arm B: T-DXd + Pembrolizumab; Arm C: Carboplatin + Paclitaxel + Pembrolizumab
Drug: Carboplatin — Standard of Care (SoC) chemotherapy by intravenous infusion
  Other Names: Carbomedac, Carbosin, Paraplatin
  Arms: Arm C: Carboplatin + Paclitaxel + Pembrolizumab
Drug: Paclitaxel — Standard of Care (SoC) chemotherapy by intravenous infusion
  Other Names: Anzatax, Ebetaxel, Oncotaxel, Paclitax, Paclitaxin, Paxene, Taxol
  Arms: Arm C: Carboplatin + Paclitaxel + Pembrolizumab
Drug: Docetaxel — Standard of Care (SoC) chemotherapy by intravenous infusion
  Other Names: Docirena, Taxceus, Taxotere
  Arms: Arm C: Carboplatin + Paclitaxel + Pembrolizumab

SUMMARY:
DESTINY-Endometrial01 will investigate the efficacy of first-line T-DXd + rilvegostomig (Arm A) and/or T-DXd+ pembrolizumab (Arm B) when compared to chemotherapy (carboplatin + paclitaxel) + pembrolizumab (Arm C), by assessment of progression free survival (PFS), as assessed by BICR, in participants with HER2-expressing (IHC 3+/2+), pMMR, primary advanced (Stage III/IV) or recurrent EC.

ELIGIBILITY:
* Key Inclusion Criteria:

  * Participants must be ≥ 18 years of age at the time of screening. Other age restrictions may apply as per local regulations.
  * Histologically confirmed diagnosis of epithelial endometrial carcinoma. All histologies are allowed except for sarcomas (carcinosarcomas are allowed).
  * Following surgery or diagnostic biopsy, participant must have primary advanced disease (Stage III/IV) or first recurrent endometrial cancer and meet at least one of the following criteria:

    * Primary Stage III (per FIGO 2023) disease with measurable disease at baseline per RECIST 1.1 based on the investigator's assessment.
    * Primary Stage IV disease (per FIGO 2023) regardless of presence of measurable disease at baseline.
    * First recurrent disease regardless of presence of measurable disease at baseline.
  * Endometrial cancer with HER2 IHC expression of 3+ or 2+ as assessed by prospective central testing.
  * Endometrial cancer that is determined pMMR by prospective central IHC testing.
  * Provision of adequate FFPE tumor tissue sample of a tumor lesion that was not previously irradiated for central HER2, MMR, and PD-L1 IHC testing and valid central test results for randomization/ stratification.
  * Prior therapy:

    * Naïve to first-line systemic anticancer therapy. Participants may have received one prior line of adjuvant/neoadjuvant chemotherapy with curative intent (chemotherapy or chemoradiation) if disease recurrence or progression occurred ≥ 6 months after last dose of chemotherapy. Prior trastuzumab in the adjuvant/neoadjuvant setting is allowed.
    * No prior exposure to ADCs or immune checkpoint inhibitors including (but not limited to) anti-PD-1/PD-L1/PD-L2 and anti-CTLA-4 antibodies and therapeutic anticancer vaccines.
    * Participants may have received prior radiation therapy for the treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy. Adequate treatment washout period is required.
  * Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
  * Left ventricular ejection fraction (LVEF) ≥ 50% within 28 days before randomization.
  * Adequate organ and bone marrow function within 14 days before randomization.
* Key Exclusion Criteria:

  * History of organ transplant
  * Uncontrolled intercurrent illness, including, but not limited to ongoing or active known infection, serious chronic gastrointestinal conditions associated with diarrhea and active non-infectious skin disease requiring systemic treatment.
  * Spinal cord compression or clinically active central nervous system metastases
  * Participants with a medical history of myocardial infarction (MI) within 6 months before randomization, or symptomatic congestive heart failure (CHF) (NYHA Class II to IV), clinically significant arrhythmia, or cardiomyopathy of any etiology. Participants with troponin levels above ULN at screening (as defined by the manufacturer), should have a cardiologic consultation before enrollment to rule out MI
  * History of (non-infectious) ILD/pneumonitis that required steroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
  * Lung criteria:

    * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within 3 months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion etc.).
    * Any autoimmune, connective tissue or inflammatory disorders where there is documented, or a suspicion of pulmonary involvement at the time of screening.
    * Prior pneumonectomy (complete).
  * Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
  * Active primary immunodeficiency/ active infectious disease(s) including:

    * Tuberculosis (TB)
    * HIV infection that is not well controlled.
    * Chronic or active hepatitis B, chronic or active hepatitis C; however, participants who have chronic hepatitis B and are receiving suppressive antiviral therapy are allowed to be enrolled if alanine aminotransferase (ALT) is normal and viral load is controlled.
  * Any concurrent anticancer treatment without an adequate washout period prior to the first dose of study intervention. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., HRT) is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-01-19 (Estimated); Study Completion 2031-02-19 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), as assessed by BICR | Until progression or death due to any cause (assessed up to approximately 45 months).
  Defined as time from randomization until progression per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR), or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until the date of death due to any cause (assessed up to approximately 70 months).
  Defined as the time from randomization until the date of death due to any cause.
Progression Free Survival (PFS) as assessed by the investigator | Until progression or death due to any cause (assessed up to approximately 70 months).
  PFS by investigator has the same attributes as estimand of PFS by BICR except tumor assessment is by the investigator.
Time from randomization to second progression or death (PFS2) | Until the earliest of the progression event (following the initial investigator-assessed progression), after first subsequent therapy, or death (assessed up to approximately 70 months).
  PFS2 will be defined as the time from randomization to the earliest of the progression event (following the initial investigator-assessed progression), after first subsequent therapy, or death.
Objective response rate (ORR), as assessed by BICR and investigator | Until progression or the starting of subsequent anticancer therapy (assessed up to approximately 45 months).
  ORR as assessed and confirmed by BICR is defined as the proportion of participants who have a complete response (CR) or partial response (PR), as determined and confirmed by BICR. ORR as assessed and confirmed by the investigator has the same attributes as estimand of ORR by BICR except tumor assessment per the investigator.
Duration of response (DoR), as assessed by BICR and investigator | Until progression or death due to any cause (assessed up to approximately 45 months).
  DoR as assessed by BICR will be defined as the time from the date of first documented response of confirmed responders until date of documented progression per RECIST 1.1, or death due to any cause.
  DoR as assessed by the investigator has the same attributes as estimand of DoR by BICR except tumor assessment per the investigator.
Safety and tolerability | Safety is assessed until the 90 days (+7) after the last dose (assessed up to approximately 70 months).
  Safety and tolerability will be evaluated in terms of AEs/serious AEs (SAEs), AESI, vital signs, clinical safety laboratory assessments, ECG and ECHO/MUGA scan results.
Pharmacokinetics of T-DXd, total anti-HER2 antibody, DXd and rilvegostomig | Up to safety follow-up period (assessed up to approximately 45 months).
  Serum concentration of T-DXd, total anti-HER2 antibody, DXd and rilvegostomig.
Immunogenicity of T- DXd and rilvegostomig | Up to safety follow-up period (assessed up to approximately 45 months).
  Presence of ADAs for T-DXd or rilvegostomig.
Patient-reported tolerability | Up to progression as assessed by BICR (assessed up to approximately 45 months).
  Patient-reported tolerability will be described among participants, as treated, using the following outcomes:
  * Symptomatic AEs: Descriptive summary of the proportion of participants reporting symptomatic AEs while on treatment, as assessed by items from the EORTC Item Library and the FACT/GOG-NTX-4
  * Overall side-effect bother: Descriptive summary of the proportion of participants reporting overall side-effect bother on the PGI-TT while on treatment
Progression-free survival (PFS) according to MMR status to determine the clinical utility of a MMR diagnostic test | Through completion of study, assessed up to approximately 70 months.
  PFS is defined as time from randomization until progression per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by BICR, or death due to any cause.
Overall survival (OS) according to MMR status to determine the clinical utility of a MMR diagnostic test | Through completion of study, assessed up to approximately 70 months.
  OS defined as the time from randomization until the date of death due to any cause.
Progression-free survival (PFS) according to HER2 expression to determine the clinical utility of a HER2 diagnostic test | Through completion of study, assessed up to approximately 70 months.
  PFS is defined as time from randomization until progression per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by BICR, or death due to any cause.
Overall survival (OS) according to HER2 expression to determine the clinical utility of a HER2 diagnostic test | Through completion of study, assessed up to approximately 70 months.
  OS is defined as the time from randomization until the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (221):
- United States (54):
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Sylmar, California
  - Research Site, Fort Myers, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Arlington Heights, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Hackensack, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Saint Johnsbury, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Australia (4):
  - Research Site, Blacktown
  - Research Site, East Melbourne
  - Research Site, Nedlands
  - Research Site, South Brisbane
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
  - Research Site, Wein
- Belgium (6):
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Goiânia
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Teresina
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (27):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yibin
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Odense
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- France (12):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Plérin
  - Research Site, Poitiers
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
- Germany (12):
  - Research Site, Berlin
  - Research Site, Chemnitz
  - Research Site, Dessau
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Münster
  - Research Site, Saarbrücken
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- Italy (10):
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Torino
  - Research Site, Turin
- Japan (20):
  - Research Site, Akashi-shi
  - Research Site, Ginowan-shi
  - Research Site, Hidaka-shi
  - Research Site, Isehara-shi
  - Research Site, Kashiwa
  - Research Site, Kashiwa-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Morioka
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Tokyo
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Norway (2):
  - Research Site, Oslo
  - Research Site, Stavanger
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Siedlce
  - Research Site, Szczecin
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, El Palmar
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (4):
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala
- Switzerland (4):
  - Research Site, Frauenfeld
  - Research Site, Liestal
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (7):
  - Research Site, Bath
  - Research Site, Cambridge
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/